CLINICAL TRIAL: NCT02817685
Title: Follow-up Strategy of Chronic Hepatitis B for Early Detection and Diagnosis of Hepatocellular Carcinoma: A Randomized Control Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Rongqin Zheng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: SYSU2016
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Hepatitis B
Keywords: surveillance; hepatocellular carcinoma; ultrasound; cirrhosis; chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Carcinoma, Hepatocellular; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 1: Chronic Hepatitis B patient
  Interventions: Other: 3 months
- 2: Chronic Hepatitis B patient
  Interventions: Other: 6 months
- 3: cirrhotic patient
  Interventions: Other: 3 months
- 4: cirrhotic patient
  Interventions: Other: 6 months
- 5: ultrasound-difficult patient
  Interventions: Other: 3 month ultrasound(US)+3 month CT/MRI+3 month US+3 month CT/MRI
- 6: ultrasound-difficult patient
  Interventions: Other: 6 months

INTERVENTIONS:
Other: 3 months
  Groups: 1; 3
Other: 6 months
  Groups: 2; 4; 6
Other: 3 month ultrasound(US)+3 month CT/MRI+3 month US+3 month CT/MRI
  Groups: 5

SUMMARY:
This study is a randomized control prospective study. The aim of this study is to establish an all-round and convenient follow-up strategy of Chronic Hepatitis B for early detection and diagnosis of Hepatocellular Carcinoma (HCC), by investigating whether different surveillance time intervals and surveillance methods are beneficial for chronic hepatitis B and cirrhotic patients with different risk of HCC.

DETAILED DESCRIPTION:
Surveillance of chronic hepatitis B and cirrhotic patients had been demonstrated to increase chances of curative treatment for hepatocellular carcinoma. However, the optimal surveillance interval for different risk patients is still controversial. The AASLD and EASL-EORTC guidelines recommend chronic hepatitis B patients undergoing ultrasound surveillance at a time interval of 6 months, but the Japanese HCC guideline recommend the very-high risk patients undergoing ultrasound surveillance at a time interval of 3 or 4 months.

The incidence of HCC is 0.3%-0.8% in the chronic hepatitis B patients and 2%-8% in cirrhotic patients, thus recalling a different follow-up strategy for different stage of chronic hepatitis B patients. Besides, ultrasound is the admitted surveillance tool for HCC for its convenience and cost-effectiveness. However, the sensitivity of ultrasound detecting HCC will remarkably decrease because of the influence of ribs, pulmonary and gastrointestinal gas, cirrhosis and fatty liver. So it is necessary to incorporate computed tomography (CT) or magnetic resonance imaging (MRI) into the follow-up strategy of very high risk patient such as patients with cirrhosis or history of HCC.

The aim of this study is to investigate whether different surveillance time intervals and surveillance methods are beneficial for chronic hepatitis B and cirrhotic patients with different risk of HCC, ultimately establish an all-round and convenient follow-up strategy of Chronic Hepatitis B for early detection and diagnosis of HCC.

ELIGIBILITY:
Inclusion Criteria:

1. HBV-Ag positive( >6 months)
2. age among 18 and 80 years

Exclusion Criteria:

1. patients with hepatocellular carcinoma
2. patients were diagnosis hepatocellular carcinoma within 3 months of inclusion;
3. patients with alcoholic hepatitis or autoimmune hepatitis
4. patients with severe uncontrolled disease resulting in estimated life expectance less than 1 year
5. coinfection with human immunodeficiency virus(HIV)
6. cannot undergo contrast-enhanced imaging
7. refuse attending the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Hepatitis B patients
Sampling Method: Non-Probability Sample
Enrollment: 7660 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
The incidence of Hepatocellular carcinoma | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: zhongzhen zz Su, doctor, Study Director — The department of Ultrasound, the third affiliated hospital of Sun Yat-sen University
Locations (1):
- The department of Ultrasound, the third affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No